CLINICAL TRIAL: NCT02678520
Title: Phase II Randomized Clinical Trial Comparing 3-D Conformal Radiation Therapy (RT) vs. Intensity Modulated Radiation Therapy in Post- Prostatectomy Prostate Cancer Patients
Brief Title: Clinical Trial Comparing 3-D RT vs. IMRT in Post- Prostatectomy Prostate Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI no longer at institution. Study terminated prior to enrolling subjects.
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015-IIT-RT-IMRT
Record Dates: First submitted 2016-01-06; First posted 2016-02-09 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Post Operative; Radiation; Prostatectomy; 3-D CRT; IMRT; RT; CRT; Conformal Radiation Therapy; Intensity Modulated Radiation Therapy; Hormone; Surgery; Hormonal Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; bicalutamide; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3-D conformal radiation therapy (Experimental): Intervention: Radiation therapy delivered to a total dose of 6600 centigray (cGy) at 200 cGy/fraction (fx) once daily using a 3-D conformal radiation technique (3-D CRT). The volume of radiation will encompass the prostatic fossa / surgical bed including any suspected regions of microscopic disease such as positive margins, extracapsular extension and/or seminal vesicle involvement. Hormonal therapy will be required for patients with "high risk" disease (both the adjuvant and salvage groups). For patients with "low risk" disease, hormonal therapy will be as per standard of care. Hormonal therapy will typically begin 2 months prior to radiation and continue for a total of 6 months. Hormonal therapy regimen will consist of Casodex (50 mg/day po for 6 months) and Zoladex (10.8 mg sc once every 3 months x 2 injections) or Lupron (22.5 mg im once every 3 months x 2 injections) to start on day 1 once the subject has been enrolled to the clinical trial.
  Interventions: Radiation: 3-D Conformal Radiation Therapy; Drug: Casodex, Zoladex , Lupron
- Intensity modulated radiation therapy (Active Comparator): Intervention: Radiation therapy delivered to a total dose of 6600 centigray (cGy) at 200 cGy/fraction (fx) once daily using intensity modulated radiation therapy (IMRT). The volume of radiation will encompass the prostatic fossa / surgical bed including any suspected regions of microscopic disease such as positive margins, extracapsular extension and/or seminal vesicle involvement. Hormonal therapy will be required for patients with "high risk" disease (both the adjuvant and salvage groups). For patients with "low risk" disease, hormonal therapy will be as per standard of care. Hormonal therapy will typically begin 2 months prior to radiation and continue for a total of 6 months. Hormonal therapy regimen will consist of Casodex (50 mg/day po for 6 months) and Zoladex (10.8 mg sc once every 3 months x 2 injections) or Lupron (22.5 mg im once every 3 months x 2 injections) to start on day 1 once the subject has been enrolled to the clinical trial.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Casodex, Zoladex , Lupron

INTERVENTIONS:
Radiation: 3-D Conformal Radiation Therapy — Radiation delivered after surgery to remove the prostate, using 3-D Conformal Radiation Therapy. Radiation will be delivered to prostatic fossa / surgical bed including any suspected regions of microscopic disease such as positive margins, extracapsular extension and/or seminal vesicle involvement.
  The total dose of radiation will be 6600 centigray (cGy) at 200 cGy/fraction (fx) given once daily .
  Other Names: 3-D CRT
  Arms: 3-D conformal radiation therapy
Radiation: Intensity Modulated Radiation Therapy — Radiation delivered after surgery to remove the prostate, using Intensity Modulated Radiation Therapy. Radiation will be delivered to prostatic fossa / surgical bed including any suspected regions of microscopic disease such as positive margins, extracapsular extension and/or seminal vesicle involvement.
  The total dose of radiation will be 6600 centigray (cGy) at 200 cGy/fraction (fx) given once daily .
  Other Names: IMRT
  Arms: Intensity modulated radiation therapy
Drug: Casodex, Zoladex , Lupron — Hormonal Therapy (6 Months): Required for "High Risk" Groups, and as per Standard of Care for "Low Risk" Groups.
  Hormonal therapy protocol regimen for the high risk "adjuvant" and "salvage" groups will consist of Casodex (50 mg/day po for 6 months) and Zoladex (10.8 mg subcutaneously once every 3 months x 2) or Lupron (22.5 mg given intramuscularly once every 3 months x 2 injections or 7.5 mg IM q once monthly x 6) to start on day 1 of the clinical trial.
  Hormonal therapy will typically begin 2 months prior to radiation and continue for a total of 6 months.
  Other Names: Hormone Therapy

SUMMARY:
Compare the incidence of acute rectal, bladder and other acute toxicities between 3-D Conformal Radiation Therapy (RT/CRT) and Intensity Modulated Radiation Therapy (IMRT) in Post-Prostatectomy Prostate Cancer Patients treated with post-operative radiation therapy

DETAILED DESCRIPTION:
In 2015, the American Cancer Society estimates that almost 220,800 men are expected to be diagnosed with prostate cancer, and about 27,540 men are expected to die of this disease. Curative treatment of prostate cancer consists of either surgery (i.e., radical prostatectomy) or radiation therapy (RT). Approximately one-third of men who undergo a prostatectomy will require post-operative adjuvant or salvage RT.

During the last 2 decades, the techniques used to deliver RT have evolved from 2-D RT in the 1980's and early 1990's, to 3-D conformal RT (3-D CRT) in the late 1990's, to intensity modulated radiation therapy (IMRT) within the last decade.

To date, no randomized prospective head to head comparison between 3-D CRT and IMRT to assess toxicity differences has ever been conducted in the treatment of post-prostatectomy prostate cancer patients. Retrospective evidence suggests comparable acute and late genitourinary (GU) and gastrointestinal (GI) toxicity. In addition, no postoperative randomized trials investigating hormonal therapy (HT) and RT have been published, but three prior phase III studies of men treated definitively for prostate cancer, one by the Radiation Therapy Oncology Group (RTOG) (86-10), one by investigators at Harvard, and one by the Trans-Tasman Radiation Oncology Group, concluded that neoadjuvant and concurrent short-term hormonal therapy (i.e., 4-6 months) RT reduces cause-specific mortality compared with RT alone.

The purpose of this study is to estimate, correlate, and compare the incidence of acute rectal, bladder and other acute toxicities between 3-D CRT and IMRT in prostate cancer patients treated with post-operative radiation therapy, to quantify, compare, and correlate the dose volume histogram (DVH) doses (e.g., Vmean, Vmedian, V25, V50, V75) to the surrounding critical organs (i.e., rectum and bladder) between 3-D CRT and IMRT, and to measure, compare, and correlate the quality of life scores of participants using the EORTC Quality of Live Questionnaires (QLQ), called "QLQ-C30" and "EPIC-26". These survey instruments will measure quality of life differences during the study; the comparison will be done between 3-D CRT and IMRT treatment arms.

Hormonal therapy will also be required for patients with high risk disease (both the adjuvant and salvage groups) and as per standard of care for patients with low risk disease, but is not explored in this study.

There are 2 arms (groups) in this study:

Arm 1: 3-D Conformal Radiation Therapy (plus hormonal therapy)

Arm 2: Intensity Modulated Radiation Therapy (plus hormonal therapy)

ELIGIBILITY:
INCLUSION Criteria:

Subjects must meet all of the inclusion criteria to participate in this study.

* Histologically documented adenocarcinoma of the prostate.
* Status post radical prostatectomy with sampling of the pelvic lymph nodes with histologically confirmed adenocarcinoma of the prostate, with the patients falling into either the "adjuvant low or high risk groups" or the "salvage low or high risk groups" as indicated below. In those cases where patients undergo a prostatectomy without any sampling of the pelvic lymph nodes, patients will be also considered eligible if they are found to have a negative pelvic CT or MRI scan which shows no evidence of lymphatic nodal metastases after the prostatectomy.

  * "Adjuvant High Risk Group" are those patients with an undetectable or persistent/decreasing PSA levels (before starting therapy) who MUST be able to start radiation therapy treatments within 6 months of radical prostatectomy with at least ONE of the 3 disease features:

    * Pathologic T2N0 (with no clinical evidence of metastases) and Gleason Score ≥ 8
    * Pathologic T3aN0 (with no clinical evidence of metastases) with Extra-Capsular Extension and Gleason Score ≥ 8
    * Pathologic T3bN0 (with no clinical evidence of metastases) with any Gleason Score
  * "Salvage High Risk Group" are those patients who experience a PSA failure (defined as at least 1 detectable PSA level > 0.2 ng/ml or at least 2 consecutive increases in PSA levels over baseline which are at least 1 month apart after radical prostatectomy) with at least ONE of the 4 following features:

    * Pathologic T3bN0 disease (with no clinical evidence of metastases),
    * Pathologic T2-3aN0 disease (with no clinical evidence of metastases) with Gleason Score ≥ 8,
    * Pathologic T2-3aN0 disease (with no clinical evidence of metastases) with PSA Doubling Time ≤ 10 months,
    * Pathologic T2-3aN0disease (with no clinical evidence of metastases) with Pre-RT PSA level ≥ 1.0 ng/ml
  * "Adjuvant Low Risk Group" are those patients with an undetectable or persistent/decreasing PSA levels (before starting therapy) who MUST be able to start radiation therapy treatments within 6 months of radical prostatectomy with at least ONE of the 2 disease features:

    * Pathologic T2N0 (with no clinical evidence of metastases), Gleason Score ≤ 7, with positive margins
    * Pathologic T3aN0 (with no clinical evidence of metastases) with Extra-Capsular Extension, Gleason Score ≤ 7, with or without positive margins
  * "Salvage Low Risk Group" are those patients who experience a PSA failure (defined as at least 1 detectable PSA level > 0.2 ng/ml or at least 2 consecutive increases in PSA levels over baseline which are at least 1 month apart after radical prostatectomy) with the following feature: - Pathologic T2-3aN0 disease (with no clinical evidence of metastases) with Gleason Score ≤7, with or without positive margins
* Neoadjuvant hormonal therapy prior to radical prostatectomy is allowed, and post-prostatectomy hormonal therapy prior to any protocol therapy is also allowed.
* Prior chemotherapy, and/or radiation therapy is allowed if it has been at least 3 years or longer since those therapies were given from the time of registration, with the exception of previous pelvic radiation which is NOT allowed under any circumstances.
* Karnofsky Performance Status ≥ 70. (Appendix A)
* Hematologic parameters must be within the following limits:

  * WBC ≥ 3,000/uL
  * Platelet Count ≥ 100,000/uL
  * Hemoglobin level ≥ 10.0 g/dl
* Patients with a history of an invasive malignancy within the last 3 years are not eligible for the protocol; patients who are NED from a prior invasive malignancy for at least 3 years or longer are eligible for the trial. Patients with history of benign tumors such as a pituitary macroadenomas, meningiomas, or craniopharyngiomas are eligible as long as the benign tumor is under local control regardless of the time frame. Patients with concurrent adequately treated basal cell or squamous cell carcinoma of the skin are also eligible for the protocol.
* Patients must sign an Informed Consent Form.
* Must not have concomitant medical, psychological or social circumstances which would interfere with compliance with the protocol treatment and follow-up.
* Age ≥ 18 years.
* Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter, which should be for at least 6 months after the completion of protocol therapy.

EXCLUSION CRITERIA

Subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.

* Patients who have received prior pelvic irradiation are not eligible.
* Any coexisting medical condition precluding full compliance with the study.
* Patients with active infections or known infection with HIV. Testing for HIV status will not be required.
* Psychological, familiar, sociological or geographical conditions which would not permit compliance with the study protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Acute rectal, bladder and other toxicity rates - For participants 1 through 10 in each treatment arm | Toxicity measured weekly starting at pre-treatment eval. and ending at end of treatment of participant 10 in both arms (Btwn approx. 7 to 11 wks per participant/through end of study; approx. 2 years)
  Acute rectal, bladder and other toxicity rates will be estimated and 95% exact binomial confidence intervals will be calculated. Toxicity will be measured via analysis of patient adverse events (physiological parameter). Adverse events will be scored using NCI Common Toxicity Criteria for Adverse Events v 4.0.3 (June 14, 2010). A two-sample binomial test will be used. This time point is an interim toxicity monitoring event designed to protect against the unlikely event of significantly more grade 2 or higher toxicities in one treatment vs. the other. If at any point, after the first 10 patients in each arm, the grade 2 or higher acute toxicity rate in either arm is more than double the grade 2 or higher acute toxicity rate in the other treatment arm, enrollment will be suspended and review of safety profiles conducted. The PI and Data Safety Monitoring Committee will then either modify the protocol or close the study to accrual.
Acute rectal, bladder and other toxicity rates - For all 100 study participants | Toxicity measured weekly starting at pre-treatment eval. and ending at end of treatment of participant 100 (Btwn approx. 7 to 11 wks per participant/through end of study; approx. 2 years)
  After safety issues, if any, have been resolved and study continued, the TOTAL of ALL 100 subjects (50 in each treatment arm) will be measured thus: Acute rectal, bladder and other toxicity rates will be estimated and 95% exact binomial confidence intervals will be calculated. To compare these rates between 3-D CRT and IMRT treatment arms, a two-sample binomial test will be used. Toxicity will be measured via analysis of patient adverse events (physiological parameter). Adverse events will be scored using NCI Common Toxicity Criteria for Adverse Events v 4.0.3 (June 14, 2010).
Dose Volume Histogram (DVH) dose quantification and comparison | DVH assessed at end of radiation therapy for each participant (Btwn approx. 7 to 11 wks for each participant) Overall DVH values compared at end of study-approx. 2 years)
  To quantify and compare the dose volume histogram (DVH) doses (e.g., Vmean, Vmedian, V25, V50, V75) to the surrounding critical organs (i.e., rectum and bladder) between 3-D CRT and IMRT, a two-sample t-test will be used.
Quality of Life measure and comparison - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ C-30) | EORTC QLQ C-30 will be assessed 2 times during each participant's study enrollment: at pre-treatment eval. (Wk 0), + after completion of radiation therapy (Betwn approx. wks 7 to 11) Overall scores will be compared at end of study - approx. 2 years
  To measure and compare participants' quality of life, overall scores will be obtained from participants via the EORTC QLQ C-30 survey instrument. This tool is used for each participant's measure of their own quality of life with this cancer. A two-sample t-test will then be used to make the comparison between treatment arms.
Quality of Life measure and comparison - Expanded Prostate Cancer Index Composite 26 (EPIC-26) | EPIC-26 will be assessed 2 times during each participant's study enrollment: at pre-treatment eval. (Wk 0), + after completion of radiation therapy (Betwn approx. wks 7 to 11) Overall scores will be compared at end of study - approx. 2 years
  To measure and compare participants' quality of life, overall scores will be obtained from participants via the EPIC-26 survey instrument. This tool is used for each participant's measure of their own quality of life with this cancer. A two-sample t-test will then be used to make the comparison between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Parvesh Kumar, MD, Principal Investigator — University of Kansas Medical Center - Cancer Center
Locations (1):
- The University of Kansas Cancer Center (KUCC), Fairway, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pilepich MV, Winter K, John MJ, Mesic JB, Sause W, Rubin P, Lawton C, Machtay M, Grignon D. Phase III radiation therapy oncology group (RTOG) trial 86-10 of androgen deprivation adjuvant to definitive radiotherapy in locally advanced carcinoma of the prostate. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1243-52. doi: 10.1016/s0360-3016(01)01579-6. PMID 11483335
- [Background] D'Amico AV, Manola J, Loffredo M, Renshaw AA, DellaCroce A, Kantoff PW. 6-month androgen suppression plus radiation therapy vs radiation therapy alone for patients with clinically localized prostate cancer: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):821-7. doi: 10.1001/jama.292.7.821. PMID 15315996
- [Background] Denham JW, Steigler A, Lamb DS, Joseph D, Mameghan H, Turner S, Matthews J, Franklin I, Atkinson C, North J, Poulsen M, Christie D, Spry NA, Tai KH, Wynne C, Duchesne G, Kovacev O, D'Este C; Trans-Tasman Radiation Oncology Group. Short-term androgen deprivation and radiotherapy for locally advanced prostate cancer: results from the Trans-Tasman Radiation Oncology Group 96.01 randomised controlled trial. Lancet Oncol. 2005 Nov;6(11):841-50. doi: 10.1016/S1470-2045(05)70348-X. PMID 16257791
- See also: American Cancer Society, Cancer Facts and Figures, 2014, p. 4 — http://www.cancer.org/acs/groups/content/@research/documents/webcontent/acspc-042151.pdf